CLINICAL TRIAL: NCT03881631
Title: Mindfulness-Based Stress Reduction for Family Caregivers of Dementia Patients
Brief Title: Improving Well-Being for Older Adult Family Dementia Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Kathi Heffner, Associate Professor, University of Rochester
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00000881; R01AG052495 (NIH)
Record Dates: First submitted 2019-03-15; First posted 2019-03-19 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Stress, Psychological
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness Based Stress Reduction (MBSR) Program (Experimental): The MBSR program is an eight-week-long course designed to teach subjects how to develop their inner resources in the service of taking better care of themselves. MBSR training includes the learning and refining of a range of skills aimed at increasing relaxation and awareness of physical experiences and sensations related to physical symptoms, emotions, and thoughts. Special emphasis is placed on movement, meditation, and breathing.
  Interventions: Behavioral: Mindfulness Based Stress Reduction Program
- Living Well (LW) Program (Active Comparator): LW is an eight-week course of group presentations and discussions on topics related to the promotion of health and well-being in the context of dementia caregiving. LW is designed to teach participants how to improve their physical and emotional health as a complement to traditional medical treatments.
  Interventions: Behavioral: Living Well Program
- Usual Care (No Intervention): The usual care arm is a no intervention group wherein participants experience their usual circumstances.

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction Program — Group-based intervention
  Other Names: MBSR
  Arms: Mindfulness Based Stress Reduction (MBSR) Program
Behavioral: Living Well Program — Group-based intervention
  Arms: Living Well (LW) Program

SUMMARY:
This study will examine the effects of the Mindfulness-Based Stress Reduction (MBSR) program and the Living Well program, compared to a control group, to see if the programs might be associated with better immune function (response to current influenza vaccine), physical and emotional health, and well-being.

DETAILED DESCRIPTION:
A considerable literature documents that a wide variety of psychosocial interventions can lessen the psychological burden of family or spousal dementia caregiving. Some caregiver intervention studies have included measures of self-reported physical health and sleep, and others have focused on improving inflammation in caregivers. The current study will add to this literature by examining the effects of two behavioral interventions on adaptive immune responses, particularly, antibody response to influenza vaccination, in older adult family caregivers.

ELIGIBILITY:
Inclusion Criteria:

* 55 years of age and older
* English-speaking (consent process and assessments will be conducted in English only)
* Currently living with or in proximity to, and the primary caregiver for, a loved one with dementia who lives in the community-for the purposes of this study, "loved one" refers to a family member such as a spouse, ex-spouse, significant other, sibling, in-law, parent, or other type of close established relationship (e.g., close friend) regarded as family; "primary caregivers" provide daily informal (non-paid) in-person care.
* Currently experiencing moderate to high levels of perceived stress (PSS-10 ≥ 12) and/or caregiver burden (MCSI ≥ 5)
* Participants will be asked to stabilize medications prior to beginning the trial, and for the duration of the trial (If medication dose changes do occur, analytic models will include those changes as time-varying covariates)

Exclusion Criteria:

* Loved one with dementia currently resides in a long-term care facility (e.g., nursing home) without the caregiver.
* Given the didactic and self-directed nature of the MBSR program, individuals with major, uncorrected sensory impairments and cognitive deficits, as determined by a Montreal Cognitive Assessment (MoCA) score of 23 or lower 29, will be excluded, as will participants with other neuropsychological deficits deemed significant enough to interfere with study participation. Low literacy is not an exclusion criterion; questionnaires will be orally administered when necessary.
* Modules from the Mini International Neuropsychiatric Exam (MINI 30) will be used to exclude subjects who have these psychiatric conditions: current alcohol dependence, current non-alcohol psychoactive substance use dependence, psychotic disorders (current and lifetime), bipolar disorder, and current mood disorder with psychotic features.
* Subjects will also be excluded for the following reasons: having completed an MBSR program in the past; allergy to eggs (the influenza vaccine is most commonly manufactured using an egg-based process); history of Guillain-Barré syndrome; immunodeficiency or receipt of immunosuppressive therapy; recent major surgery; and active neoplastic disease.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2016-07-18 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
Antibody response to influenza vaccination | pre-vaccination to 6 weeks and 6 months post-vaccination
  Change in amount of antibody titers following influenza vaccination

SECONDARY OUTCOMES:
Granzyme B (GrzB) activity after influenza vaccination | pre-vaccination to 6 weeks and 6 months post-vaccination
  Change in GrzB activity, a measure of antigen-specific cytotoxic T cell activity, following influenza vaccination
Ratio of T-cell cytokines, interferon (IFN)-gamma and IL-10 | pre-vaccination to 6 weeks and 6 months post-vaccination
  Change in IFN:IL-10 ratio following influenza vaccination
Inflammatory cytokines, interleukin (IL)-6 and tumor necrosis factor (TNF)-alpha | baseline to 6 weeks to 6 months post-intervention
  Change in inflammatory cytokine levels over time

CONTACTS AND LOCATIONS:
Overall Officials: Kathi L Heffner, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing is in accordance with NIH Data Sharing Policy.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 12 months of study end

DOCUMENTS (1):
  • Informed Consent Form (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/31/NCT03881631/ICF_000.pdf